CLINICAL TRIAL: NCT00552955
Title: Effect of Fasting on the Size of Lymphangioleiomyomas in Patients With Lymphangioleiomyomatosis
Brief Title: Effect of Fasting on the Size of Abdominal Lymphatic Tumors in Women
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080016; 08-H-0016
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2016-03-21

CONDITIONS: Lymphangioleiomyomas; Tuberous Sclerosis; Lymphangioleiomyomatosis
Keywords: Lymphangioleiomyomatosis; Abdominal Lymphangioleiomyomas; Chyle; Ascites; Tuberous Sclerosis Complex; LAM
MeSH Terms: conditions — Lymphangiomyoma; Tuberous Sclerosis; Lymphangioleiomyomatosis; Ascites

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will examine the effect of fasting on lymphangioleiomyomas abdominal tumors formed from enlarged lymph nodes containing lymphatic fluid. Previous studies have determined that these tumors increase in size in the evening, but this result could stem from the fact that previous study participants were tested after eating lunch. The purpose of the study is to help researchers understand the factors that produce changes in size of lymphangioleiomyomas, as well as to improve the ability of medical professionals to diagnose lymphangioleiomyomas and avoid confusing these tumors with other malignant tumors.

Volunteers must be women who are at least 18 years of age and who have been diagnosed with lymphangioleiomyomas in the abdominal or pelvic areas. Candidates who have had lung or kidney transplants or who have type 1 diabetes will be excluded. Candidates will be screened with a physical examination and medical history.

During the study, participants will be admitted to a National Institutes of Health clinical center for three days to undergo a number of tests. Tests will include routine blood and urine tests, and electrocardiogram, research blood testing, and abdominal and pelvic ultrasounds....

DETAILED DESCRIPTION:
Lymphangioleiomyomatosis (LAM) is a rare disease of women that is characterized by a proliferation of abnormal smooth muscle-like cells (LAM cells) in the lungs, which leads to cystic destruction of the lung parenchyma, in the axial lymphatics, resulting in lymphangioleiomyomas, and in abdominal angiomyolipomas, primarily in the kidneys. Lymphangioleiomyomas may cause abdominal distension and compress abdominal organs, producing obstipation, bladder obstruction and neurological deficits. Leakage of chyle may be responsible for ascites and pleural effusions. The lymphangioleiomyomas may change in size during the day. This variation in tumor size may be due to increased chyle formation or alterations in lymphatic flow. These studies however, were not performed with research subjects who were fasting. Our hypothesis is that the ingestion of food increases chyle formation and lymphatic flow, which in turn increases the size of the lymphangioleiomyomas. The aim of this study is to test this hypothesis. We propose to conduct a study in 30 LAM patients who have lymphangioleiomyomas to determine whether the ingestion of food, by increasing chyle formation and lymphatic flow, increases the size of the lymphangioleiomyomas.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals who are 18 years of age or older with any of the following:

1. Lymphangioleiomyomatosis
2. Abdominal or pelvic lymphangioleiomyomas equal to or greater than one centimeter in diameter in the non-fasting state.

EXCLUSION CRITERIA:

Individuals with any of the following:

1. Lung transplantation
2. Kidney transplantation
3. Lymphangioleiomyomas smaller than one centimeter in diameter in the non-fasting state.
4. Pregnancy or lactation.
5. Type 1 diabetes.
6. Inability to give informed consent.
7. Currently taking rapamycin.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-10-26; Study Completion 2016-03-21

CONTACTS AND LOCATIONS:
Overall Officials: Angelo M Taveira-DaSilva, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kitaichi M, Nishimura K, Itoh H, Izumi T. Pulmonary lymphangioleiomyomatosis: a report of 46 patients including a clinicopathologic study of prognostic factors. Am J Respir Crit Care Med. 1995 Feb;151(2 Pt 1):527-33. doi: 10.1164/ajrccm.151.2.7842216.
- [Background] Chu SC, Horiba K, Usuki J, Avila NA, Chen CC, Travis WD, Ferrans VJ, Moss J. Comprehensive evaluation of 35 patients with lymphangioleiomyomatosis. Chest. 1999 Apr;115(4):1041-52. doi: 10.1378/chest.115.4.1041. PMID 10208206
- [Background] Johnson SR, Tattersfield AE. Clinical experience of lymphangioleiomyomatosis in the UK. Thorax. 2000 Dec;55(12):1052-7. doi: 10.1136/thorax.55.12.1052. PMID 11083892